CLINICAL TRIAL: NCT03670381
Title: Investigation of the HDAC4 Copy Number Variation and Its Effect on Gene and Protein Expression in Patients With ASD
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201608089RIN
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Ten mL of peripheral blood will be drawn for DNA and cell line preparation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASD group: ASD patients with HDAC4 CNVs
  Interventions: Other: Psychiatric diagnosis
- TD group: Typically developing controls without lifetime ASD or a family history of ASD
  Interventions: Other: Psychiatric diagnosis

INTERVENTIONS:
Other: Psychiatric diagnosis

SUMMARY:
Specific Aims of this study:

1. To understand the distribution of HDAC4 CNV in the families of the ASD patients with HDAC4 CNV;
2. To perform the analysis of gene expression;
3. To investigate the HDAC4 protein level expression;
4. To investigate the correlation of clinical/cognitive features with HDAC4 CNV, RNA and protein expression in ASD patients, and compare with their unaffected family members.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a common neurodevelopmental disorder affecting up to 1/50 in the world and 1% in Taiwan. ASD is a clinically and genetically heterogeneous complex disorder with high heritability. Due to its high prevalence, lifetime impairment and no effective prevention and treatment, ASD has been prioritized for molecular genetic study. Among the genetic findings based on our copy number variation (CNV) analysis of 335 patients with ASD, HDAC4 gene is selected to help us understand the pathogenesis of ASD by investigating parent-of-origin and the gene and protein expression of this gene, alongside neurocognitive and behavioral phenotypes.

Based on our findings on HDAC4 CNV analysis, the patients with HDAC4 CNVs (~30 patients) and their families will be invited to participate the investigation of the CNV, RNA and protein expression analysis. Five healthy controls without any diagnosis of psychiatric disorders will be recruited to perform the comparison with ASD patients with HDSC4. The autistic symptoms and behavioral phenotypes assessed by the Chinese SCQ and SRS, and the cognitive function assessed by intelligence test and WCST will be used to reveal the associations among the CNVs, RNA expression, protein level and clinical/cognitive phenotypes.

According to our previous CNV findings at the HDAC4 locus, we expect to find CNV in HDAC4 variation in another independent sample of our ASD cohort and to explore how HDAC4 CNVs affect the RNA and protein expression of HDAC4. We anticipate our endeavors will provide the comprehensive profiles of the CNV, RNA and protein expressions and the clinical features of ASD patients with HDAC4 CNVs and contribute to our understanding of the pathogenesis of ASD.

ELIGIBILITY:
Inclusion Criteria:

* ASD group: Subjects who met the diagnostic criteria of either autistic disorder or Asperger's disorder defined by the DSM-IV criteria.

Exclusion Criteria:

* TD group: Subjects with any current or lifetime DSM-IV psychiatric disorders.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 30 ASD patients with HDAC4 CNVs and 5 healthy controls without any diagnosis of psychiatric disorders will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Copy number variation (CNV) analysis | 5 days
  Using SYBR-Green based real-time qPCR (Applied Biosystems, Forster, CA) to detect the CNVs encompassing HDAC4 gene in participants.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan